CLINICAL TRIAL: NCT03497039
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Arm, Steady-State Pharmacokinetic and Disposition Study Characterizing Diclofenac's Plasma and Knee Exposure in Osteoarthritis (OA) Subjects Undergoing Scheduled Arthroplasty After Treatment With Diclofenac Diethylamine (DDEA) 2.32% Gel
Brief Title: A Study to Characterize Diclofenac's Plasma and Knee Exposure After Application of Diclofenac Gel to the Knee of Subjects With Osteoarthritis That Have a Scheduled Arthroplasty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 208901
Record Dates: First submitted 2018-04-05; First posted 2018-04-13 (Actual); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — diclofenac diethylamine; di-N-desethylamiodarone; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental): In the active treatment arm, DDEA gel will be applied topically at a dose of 4 gram (g) on 400 square centimeter (cm^2) twice a day for 7 days to the target knee (the knee planned for arthroplasty surgery).
  Interventions: Drug: Diclofenac Diethylamine (DDEA) gel
- Placebo Control (Placebo Comparator): In the placebo control arm, placebo gel will be applied topically at a dose of 4 gram (g) on 400 square centimeter (cm^2) twice a day for 7 days to the target knee (the knee planned for arthroplasty surgery).
  Interventions: Other: Placebo gel

INTERVENTIONS:
Drug: Diclofenac Diethylamine (DDEA) gel — Diclofenac Diethylamine (DDEA) gel consists of 2.32% DDEA. DDEA gel will be applied twice a day for 7 days topically first and last dose by trained nurse (or designee) at study site and doses in between by a trained nurse at participant's home or other convenient location. Participants will be admitted on the day before the scheduled surgery (Day 7). The last dose of study treatment will be administered at the study site 12 hours (window -1/+3 hrs) prior to arthroplasty surgery.If surgery is delayed by up to 7 days dosing with DDEA gel twice daily can continue up to 14 days. If the surgery is delayed by more than 7 days, the participant should be withdrawn from the study.
  Arms: Active Treatment
Other: Placebo gel — Placebo gel will be applied twice a day for 7 days topically first and last dose by trained nurse (or designee) at study site and doses in between by a trained nurse at participant's home or other convenient location. Participants will be admitted on the day before the scheduled surgery (Day 7). The last dose of placebo gel will be administered at the study site 12 hours (window -1/+3 hrs) prior to arthroplasty surgery. If surgery is delayed by up to 7 days dosing with placebo gel twice daily can continue up to 14 days. If the surgery is delayed by more than 7 days, the participant should be withdrawn from the study.
  Arms: Placebo Control

SUMMARY:
The purpose of this study is to evaluate the exposure of diclofenac in the plasma and in the knee joint following topical administration of DDEA gel 4 gram (g) applied twice daily for 7 days.

DETAILED DESCRIPTION:
The study will be performed in Participants diagnosed with OA of the knee who are scheduled for arthroplasty of the knee as a treatment for their OA.

Approximately fifty (50) male and female OA participants, who, at the time of screening, are ≥50 years old, will be randomized in a 2:1 ratio: two thirds will receive DDEA gel treatment and one third placebo gel.After providing informed consent to participate in the study the participants will need to forego any non-steroidal anti inflammatory drug (NSAID) or cyclooxygenase (COX)-2 treatment for at least 7 days prior to starting study treatment (Visit 2) to allow wash-out of existing therapy and thus avoiding confounding the effect of the study treatments.

There will be 4 study center visits as follows:

Visit 1 Screening visit: Day -7 (Window: Day-10 to Day-7) Visit 2 Baseline (randomization) visit: Morning of Day 1 Visit 3 Hospital admittance through to surgery and post-surgery: Evening of Day 7 through Day 8 (Surgery may be delayed by up to 7 days) Visit 4 Final visit: Day 8 to Day 10 (Between recovery and discharge)

The Participants will be provided paracetamol as rescue medication, to be used up to a total daily dose of 4 gram (g). Rescue medication will be available from the Screening Visit (Day -7) through to end of Day 7. Should the need arise for additional pain relief, the investigators will be allowed to prescribe codeine or tramadol. Postoperative analgesia will be handled according to the surgical center's pain management procedures.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Male and female participants who, at the time of screening, are ≥ 50 years of age.
* Participant has a diagnosis of OA of the knee requiring arthroplasty and is scheduled for single knee arthroplasty, with radiographic evidence within last 6 months confirming Kellgren Lawrence grade of 2 or more.
* Participant is in general good physical health and deemed fit for surgery, as judged by the investigator and no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, respiratory rate and temperature measurement, 12 lead ECG or clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to less than 40 kg/m2; and a total body weight >50 kg (110 lbs).
* Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Female participants of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for at least 21 days after the last dose of assigned treatment. Female participants who are not of childbearing potential must meet following requirements: Female participants who are of childbearing potential and are sexually active and at risk for pregnancy must agree to use a highly effective method of contraception consistently and correctly for the duration of the active study period (onwards from screening) and for at least 21 days after the last dose of investigational product. The investigator or his or her designee, in consultation with the participant, will confirm that the participant has selected an appropriate method of contraception for the individual participant from the permitted list of contraception methods (see below) and instruct the participant in its consistent and correct use. Participants need to affirm that they meet the criteria for the correct use of at least 1 of the selected methods of contraception. The investigator or his or her designee will discuss with the participant the need to use highly effective contraception consistently and correctly according to the schedule of activities and document such conversation in the participant's chart. In addition, the investigator or his or her designee will instruct the participant to call immediately if the selected contraception method is discontinued or if pregnancy is known or suspected in the participant. Highly effective methods of contraception are those that, alone or in combination, result in a failure rate of less than 1% per year when used consistently and correctly (i.e., perfect use) and include the following a)Established use of oral, inserted, injected, transdermal, or implanted hormonal methods of contraception is allowed provided the participant plans to remain on the same treatment throughout the entire study and has been using that hormonal contraceptive for an adequate period of time to ensure effectiveness as deemed appropriate by the investigator, b) Correctly placed copper-containing intrauterine device (IUD), c) Male condom or female condom used with a spermicide (i.e., foam, gel, film, cream, or suppository), d) Male sterilization with absence of sperm in the post-vasectomy ejaculate e) Bilateral tubal ligation / bilateral salpingectomy or bilateral tubal occlusive procedure (provided that occlusion has been confirmed in accordance with the device's label), f)Female who meets the criteria for non-childbearing potential as described below. Female participants of non-childbearing potential must meet at least one of the following criteria: 1) Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed by a serum follicle-stimulating hormone (FSH) level confirming the post-menopausal state, 2) Have undergone a documented hysterectomy and/or bilateral oophorectomy, 3) Have medically confirmed ovarian failure.

All other female participants (including females with tubal ligations) will be considered to be of childbearing potential.

Exclusion Criteria:

* Participants who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or participants who are GSK employees directly involved in the conduct of the study.
* Participation in other studies involving investigational drug(s) within one month prior to study entry and/or during study participation.
* Acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Pregnant female participants.
* Breastfeeding female participants.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Participants in whom attacks of asthma, angioedema, urticaria, or acute rhinitis are precipitated by acetylsalicylic acid or other non-steroidal anti-inflammatory drugs (NSAIDs).
* Participants whose skin around the knee is broken, diseased or has skin wounds or open injuries.
* Unwilling or unable to comply with the following lifestyle guidelines described in the protocol or investigator instructions: a) Meals and Dietary Restrictions: No specific meal or dietary restriction is required for the study. Participants will follow the perioperative guidance with respect to meals and dietary restrictions as provided by the surgical center. Participants must abstain from all food and drink (except water) at least 4 hours prior to any safety laboratory evaluations, b)Alcohol, Caffeine and Tobacco: participants will follow the perioperative guidance with respect to alcohol and caffeine intake and use of tobacco- or nicotine containing products as provided by the surgical center, c) Activity: participants will follow the perioperative guidance with respect to activity as provided by the surgical center, d) Contraception: Female participants who are of childbearing potential and are sexually active and at risk for pregnancy must agree to use a highly effective method of contraception consistently and correctly for the duration of the active study period (onwards from screening) and for at least 21 days after the last dose of investigational product. The investigator or his or her designee, in consultation with the participant, will confirm that the participant has selected an appropriate method of contraception for the individual participant from the permitted list of contraception methods (see below) and instruct the participant in its consistent and correct use. Participants need to affirm that they meet the criteria for the correct use of at least 1 of the selected methods of contraception. The investigator or his or her designee will discuss with the participant the need to use highly effective contraception consistently and correctly according to the schedule of activities and document such conversation in the participant's chart. In addition, the investigator or his or her designee will instruct the participant to call immediately if the selected contraception method is discontinued or if pregnancy is known or suspected in the participant.

Highly effective methods of contraception are those that, alone or in combination, result in a failure rate of less than 1% per year when used consistently and correctly (i.e., perfect use) and include the following: 1) Established use of oral, inserted, injected, transdermal, or implanted hormonal methods of contraception is allowed provided the participant plans to remain on the same treatment throughout the entire study and has been using that hormonal contraceptive for an adequate period of time to ensure effectiveness as deemed appropriate by the investigator, 2) Correctly placed copper-containing intrauterine device (IUD), 3) Male condom or female condom used with a spermicide (i.e., foam, gel, film, cream, or suppository), 4) Male sterilization with absence of sperm in the post-vasectomy ejaculate, 5) Bilateral tubal ligation / bilateral salpingectomy or bilateral tubal occlusive procedure (provided that occlusion has been confirmed in accordance with the device's label), 6)Female who meets the criteria for non-childbearing potential as described below. Female participants of non-childbearing potential must meet at least one of the following criteria: a) Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed by a serum follicle-stimulating hormone (FSH) level confirming the post-menopausal state, b) Have undergone a documented hysterectomy and/or bilateral oophorectomy, c) Have medically confirmed ovarian failure.

All other female participants (including females with tubal ligations) will be considered to be of childbearing potential e) Screen Failures: Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently randomized. In order to ensure transparent reporting of screen failure participants, a minimal set of screen failure information will include screening number, date of screening, demography (gender, year of birth, age), screen failure details (e.g., withdrawal of consent), eligibility criteria, and any serious adverse events. Screening failures will be replaced in the recruitment schedule until the required number of participants are randomized. Individuals who do not meet the criteria for participation in this study (screen failure) may not be re-screened, f) Sponsor's Qualified Medical Personnel: The contact information for the sponsor's appropriately qualified medical personnel for the study is documented in the study contact list located in the supporting study documentation. The contact number can be used by investigational staff if they are seeking advice on medical questions or problems; however, it should be used only in the event that the established communication pathways between the investigational site and the study team are not available. It is therefore intended to augment, but not replace, the established communication pathways between the investigational site and the study team for advice on medical questions or problems that may arise during the study. The contact number is not intended for use by the participant directly, and if a participant calls that number, he or she will be directed back to the investigational site. To facilitate access to appropriately qualified medical personnel on study-related medical questions or problems, participants are provided with a contact card. The contact card contains, at a minimum, protocol identifiers, participant study numbers, contact information for the investigational site, and contact details in the event that the investigational site staff cannot be reached to provide advice on a medical question or problem identified from the participant's healthcare professional other than the investigator.

* Use of prescription or nonprescription drugs (unless deemed necessary by investigator), NSAIDs, COX-2 inhibitors and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study treatment and during the study. Specifically if, during the washout period or the treatment period, the participant is unwilling to avoid the use of any topical or systemic analgesic or anti-inflammatory treatments other than the study medication, the rescue medication, and if needed codeine or tramadol.
* Use of one or more of the following treatments prior to the screening visit or between screening and baseline visit: a) any topical NSAID treatment between screening and baseline visit, b) any intra-articular or peri-articular procedures or injections in either knee within the previous 3 months, c) any systemic treatment with corticosteroids within the previous 6 weeks (topical treatments with corticosteroids not related to either knee are permitted up to screening visit), d) any chondroprotectant or disease-modifying OA drugs, such as glucosamine or chondroitin sulfate, unless dose was stable over the previous month and will be maintained throughout the study, e) any systemic anti-inflammatory or analgesic drugs at screening if 5 times their elimination halftime exceeds 7 days (i.e., if half-life > 33.6 hrs), f) anticoagulants such as warfarin or heparin in the preceding week or antiaggregants within the previous month other than aspirin at stable low doses started at least one month before randomization and kept at a constant dose throughout the study or anticoagulant therapy for surgery, g) any other investigational drugs within the previous month or 5 half lives preceding the first dose of investigational product (whichever is longer).
* A positive urine drug screen during Screening (Day -7).
* Any condition possibly affecting drug absorption (e.g., gastrectomy).
* History of regular alcohol consumption exceeding 14 drinks/week (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
* Participants who have previously been enrolled in this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- GSK Investigational Site, Würzburg, Bavaria, Germany
- United Kingdom (4):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Clydebank
  - GSK Investigational Site, Leeds

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 4 sites in the United Kingdom and 1 site in Germany.
Pre-assignment Details: A total of 47 participants with osteoarthritis were enrolled out of which 46 were randomly assigned in 2 arms either to receive Diclofenac Diethylamine (DDEA) 2.32 percent (%) gel treatment or placebo gel. 1 participant withdrew consent before starting treatment.
Groups:
- Diclofenac Diethylamine (DDEA) Gel: Participants randomized to this group were instructed to apply DDEA 2.32% gel topically,4grams(g) for about 1minute over a region of approximately 400 square centimeter(cm^2)per knee, every 12hours (hrs) twice daily for 7days. First and last doses were applied by trained nurse at study site. Last dose of study treatment administered at study site 12hrs (-1/+3hrs) prior to arthroplasty surgery (Day 7). If surgery delayed by up to 7days dosing with DDEA gel twice daily continued up to 14days.If surgery delayed by more than 7days,participant withdrawn from study. Rescue medication (Paracetamol,500milligrams [mg] tablets) provided at screening visit and instructed to take only if needed 1or2 tablets repeated after at least 4hrs up to 4times daily, up to a maximum of 4g per day.
- Placebo Gel: Participants randomized to this group were instructed to apply Placebo gel topically, 4 g for about 1minute over a region of approximately 400 cm^2 per knee, every 12 hrs twice daily for 7days. First and last doses were applied by trained nurse at study site. Last dose of study treatment administered at study site 12hrs (-1/+3hrs) prior to arthroplasty surgery (Day 7). If surgery delayed by up to 7days dosing with DDEA gel twice daily continued up to 14days. If surgery delayed by more than 7days,participant withdrawn from study. Rescue medication (Paracetamol, 500 mg tablets) provided at screening visit and instructed to take only if needed 1or2 tablets repeated after at least 4hrs up to 4times daily, up to a maximum of 4g per day.
Period: Overall Study
Arm/Group | Diclofenac Diethylamine (DDEA) Gel | Placebo Gel
Started | 30 | 17
Treated | 29 | 17
Completed | 29 | 16
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were randomized and received at least one dose of investigational product.
Groups:
- Diclofenac Diethylamine (DDEA) Gel: Participants randomized to this group were instructed to apply DDEA 2.32% gel topically, 4 g for about 1minute over a region of approximately 400 cm^2 per knee, every 12 hrs twice daily for 7days. First and last doses were applied by trained nurse at study site. Last dose of study treatment administered at study site 12hrs (-1/+3hrs) prior to arthroplasty surgery (Day 7). If surgery delayed by up to 7days dosing with DDEA gel twice daily continued up to 14days. If surgery delayed by more than 7days,participant withdrawn from study. Rescue medication (Paracetamol, 500 mg tablets) provided at screening visit and instructed to take only if needed 1or2 tablets repeated after at least 4hrs up to 4times daily, up to a maximum of 4g per day.
- Total: Total of all reporting groups
Arm/Group | Diclofenac Diethylamine (DDEA) Gel | Placebo Gel | Total
Number analyzed (Participants) | 29 | 17 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (7.59) | 71.7 (8.63) | 71.2 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 14 | 8 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Diclofenac Concentration in Treated Knee Synovial Tissue After 7 Days Topical Application of Study Treatment to the Knee (12 Hours After Last Administration of Study Treatment)
Description: Synovial tissue was collected during surgery (participant's scheduled arthroplasty of the target knee on which study treatment was applied). Samples were analyzed for diclofenac levels using a validated bio analytical method in compliance with the applicable standard operating procedures of the bioanalytical laboratory. Synovial tissue diclofenac concentration was summarized by treatment group. Number of participants with diclofenac concentration values that were below the limit of quantification (LOQ) were replaced by 0 for placebo group. The geometric mean was calculated with a two-sided 95% confidence interval assuming data on the logarithmic scale were normally distributed.
Time Frame: At Day 8 (up to a maximum of Day 15 in case of surgery delay)
Population: Analyzable population consists of all participants who were randomized, received at least 1 dose of investigational product, completed surgery and had evaluable synovial tissue or synovial fluid sample. Here, number analyzed indicates participants with diclofenac tissue concentration values greater than LOQ.
Measure: Geometric Mean (95% Confidence Interval); unit: nanograms per gram (ng/g)
Arm/Group | Diclofenac Diethylamine (DDEA) Gel | Placebo Gel
Number analyzed (Participants) | 29 | 16
nanograms per gram (ng/g) | 1.573 [1.124 to 2.200] | NA [NA to NA] — Data could not be computed due to participants with zero values.

2. Primary Outcome: Diclofenac Concentration in Treated Knee Synovial Fluid After 7 Days Topical Application of Study Treatment to the Knee (12 Hours After Last Administration of Study Treatment)
Description: Synovial fluid was collected during surgery (participant's scheduled arthroplasty of the target knee on which study treatment was applied). Samples were analyzed for diclofenac levels using a validated bio analytical method in compliance with the applicable standard operating procedures of the bioanalytical laboratory. Synovial fluid diclofenac concentration was summarized by treatment group. Number of participants with diclofenac concentration values that were below the LOQ were replaced by 0 for placebo group. The geometric mean was calculated with a two-sided 95% confidence interval assuming data on the logarithmic scale were normally distributed.
Time Frame: At Day 8 (up to a maximum of Day 15 in case of surgery delay)
Population: Analyzable population consists of all participants who were randomized,received at least 1 dose of investigational product,completed surgery and had evaluable synovial tissue or synovial fluid sample.Here,number analyzed indicates participants with diclofenac fluid concentration values greater than LOQ.
Measure: Geometric Mean (95% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Arm/Group | Diclofenac Diethylamine (DDEA) Gel | Placebo Gel
Number analyzed (Participants) | 29 | 16
nanograms per milliliter (ng/mL) | 2.274 [1.874 to 2.759] | NA [NA to NA] — Data could not be computed due to some participants with zero values.

3. Secondary Outcome: Ratio Between Diclofenac Concentration in Treated Knee Synovial Tissue and Plasma After 7 Days Topical Application of Study Treatment to the Knee (12 Hours After Last Administration of Study Treatment)
Description: Synovial tissue was collected during surgery (participant's scheduled arthroplasty of the target knee on which study treatment was applied). Samples were analyzed for diclofenac levels using a validated bio analytical method in compliance with the applicable standard operating procedures of the bioanalytical laboratory. Diclofenac concentration values that were below the LOQ were replaced by 0 for placebo group. The ratio between diclofenac concentration in treated knee synovial tissue and plasma was calculated.
Time Frame: At Day 8 (up to a maximum of Day 15 in case of surgery delay)
Population: Analyzable population consists of all participants who were randomized, received at least 1 dose of investigational product, completed surgery and had evaluable synovial tissue or synovial fluid sample. Here, number analyzed indicates participants with diclofenac plasma concentration and tissue concentration values greater than LOQ.
Measure: Geometric Mean (95% Confidence Interval); unit: (ng/g)/(ng/mL)
Arm/Group | Diclofenac Diethylamine (DDEA) Gel | Placebo Gel
Number analyzed (Participants) | 29 | 16
(ng/g)/(ng/mL) | 0.320 [0.228 to 0.450] | NA [NA to NA] — Data could not be computed due to participants with zero values.

4. Secondary Outcome: Ratio Between Diclofenac Concentration in Treated Knee Synovial Fluid and Plasma After 7 Days Topical Application of Study Treatment to the Knee (12 Hours After Last Administration of Study Treatment)
Description: Synovial fluid was collected during surgery (participant's scheduled arthroplasty of the target knee on which study treatment was applied). Samples were analyzed for diclofenac levels using a validated bio analytical method in compliance with the applicable standard operating procedures of the bioanalytical laboratory. Diclofenac concentration values that were below the limit of quantification (LOQ) were replaced by 0 for placebo group. The ratio between diclofenac concentration in treated knee synovial fluid and plasma was calculated.
Time Frame: At Day 8 (up to a maximum of Day 15 in case of surgery delay)
Population: Analyzable population consists of all participants who were randomized, received at least 1 dose of investigational product, completed surgery and had evaluable synovial tissue or synovial fluid sample. Here, number analyzed indicates participants with diclofenac plasma concentration and fluid concentration values greater than LOQ.
Measure: Geometric Mean (95% Confidence Interval); unit: (ng/mL)/(ng/mL)
Arm/Group | Diclofenac Diethylamine (DDEA) Gel | Placebo Gel
Number analyzed (Participants) | 29 | 16
(ng/mL)/(ng/mL) | 0.463 [0.397 to 0.539] | NA [NA to NA] — Data could not be computed due to some participants with zero values.

ADVERSE EVENTS:
Time Frame: From start of treatment (Day 1) up to Day 10 (up to a maximum of Day 18 in case of surgery delay)
Description: Safety population included all participants who were randomized and received at least one dose of investigational product. All adverse events (AEs) were summarized by system organ class and preferred term. All treatment emergent AEs and serious AEs were collected and reported.
Arm/Group | Diclofenac Diethylamine (DDEA) Gel | Placebo Gel
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/17
Other Adverse Events (participants affected / at risk) | 16/29 | 10/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diclofenac Diethylamine (DDEA) Gel (N=29) | Placebo Gel (N=17)
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diclofenac Diethylamine (DDEA) Gel (N=29) | Placebo Gel (N=17)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 4 | 1
Eye injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursal fluid accumulation (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint warmth (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Blood pressure decreased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 2 | 1
Dizziness (Nervous system disorders) | 0 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0
Sensory loss (Nervous system disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Eye swelling (Eye disorders) | 1 | 0
Swelling (General disorders) | 1 | 0
Flour sensitivity (Immune system disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT03497039/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT03497039/SAP_001.pdf